CLINICAL TRIAL: NCT02039869
Title: Confocal Endomicroscopy for Non-Erosive Reflux Disease (CE NERD)
Acronym: CE_NERD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Could not recruit patients - modifying protocol and plan resubmission to our IRB
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Medical University of South Carolina (Other); Ochsner Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: HM20000591
Record Dates: First submitted 2013-12-20; First posted 2014-01-20 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Gastroesophageal Reflux Disease; Non Erosive Reflux Disease; Dyspepsia
Keywords: NERD; Non erosive reflux disease; functional dyspepsia; erosive esophagitis; confocal endomicroscopy; cell visio; proton pump inhibitor; sucralfate
MeSH Terms: conditions — Gastroesophageal Reflux; Non-Erosive Reflux Disease; Dyspepsia | interventions — Proton Pump Inhibitors; Omeprazole; Sucralfate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Proton Pump Inhibitor (Experimental): Patients will receive proton pump inhibitor therapy with omeprazole twice daily while we observe for improvement in reflux symptoms. We will compare the confocal endomicroscopy images in the responders to non-responders at the end of 8 weeks to determine if confocal endomicroscopy can select patient that would benefit most from proton pump inhibitor therapy.
  Interventions: Device: Confocal endomicroscopy; Drug: Proton pump inhibitor
- Sucralfate (Experimental): Patients will receive sucralfate therapy four times a day while we observe for improvement in reflux symptoms. We will compare the confocal endomicroscopy images in the responders to non-responders at the end of 8 weeks to determine if confocal endomicroscopy can select patient that would benefit most from sucralfate therapy.
  Interventions: Device: Confocal endomicroscopy; Drug: Sucralfate

INTERVENTIONS:
Device: Confocal endomicroscopy — The probe allows microscopic evaluation of tissue in real time during endoscopy.
  Other Names: CellVisio
Drug: Proton pump inhibitor — Acid suppressing medication (over the counter)
  Other Names: Omeprazole (Prilosec)
  Arms: Proton Pump Inhibitor
Drug: Sucralfate — Coating agent for damaged intestinal lining.
  Other Names: Carafate (sucralfate)
  Arms: Sucralfate

SUMMARY:
The purpose of this study is to find out if people who have non-erosive reflux disease (NERD) have changes the investigators can see with a microscope (called confocal endomicroscopy) that is used during endoscopy (a camera scope evaluation of the inside of your stomach and swallowing tube). Traditionally the investigators have used trials of acid blocking medications (PPIs), endoscopy and measurements of acid in the swallowing tube (the esophagus) to determine if the investigators think acid is causing troublesome symptoms. The medical community believes that these symptoms are due to increased spaces between the cells that make up the swallowing tube. The investigators can directly see those spaces with a new microscope that the investigators can pass through the camera scope.

Participants will be assigned to take one of two medications omeprazole and sucralfate (both approved medications for stomach symptoms) to treat their symptoms and record how well the treatment works. The investigators then will look to see if the microscope can predict which medication will work best for patients in the future. The investigators also plan to measure the acid levels in your swallowing tube and do a camera evaluation of your swallowing tube and stomach as this is standard for patients with your symptoms. The investigators will compare the results of those studies to the microscope findings.

DETAILED DESCRIPTION:
Study entry criteria:

The investigators plan to collaborate with three centers to ensure the data derived from this study is generalizable to academic centers as a whole and also to expedite patient recruitment. The centers that will participate are Virginia Commonwealth University, Ochsner Health System and the Medical University of South Carolina.

Patients over the age of 18 presenting to clinic with symptoms typical for reflux disease will be screened to determine if they wish to participate in the study. The site principal investigator will directly contact potential patients to see if they wish to participate. If they elect to participate they will be provided a copy of the informed consent 24 hours before their first contact with study personnel to allow time to review and determine if the wish to participate. All participants will sign a written informed consent.

Patients who wish to enter into the study and have signed an informed consent will complete a reflux disease questionnaire (RDQ). This questionnaire consists of 12 items assessing various aspects of reflux disease. A score of more than 12 will be required for study entry. Individual with a score less than 12 will not participate further in the study.

Standard of care for patients with gastroesophageal reflux disease (GERD) not responsive to proton pump inhibitors (PPI) is confirmatory testing with esophagogastroduodenoscopy (EGD) to evaluate for erosive esophagitis (EE) and testing for acid exposure to the lower esophagus with pH testing. For the purpose of this study the investigators will perform pH testing off acid suppressing medication. This is a standard test for determining if the patient has acid exposure to the esophagus. Typically patients are placed on twice daily (BID) PPI or sucralfate if testing reveals significant acid exposure.

Erosive esophagitis will be differentiated from NERD by endoscopic findings aided by FICE (or NBI/iScan) and magnification techniques that the investigators standardly employ in clinical practice. Patients that are found to have EE will not participate further in the study and will be treated appropriately for their illness with increased acid suppression. Patients without EE at the time of endoscopy will be enrolled for study as presumed cases of NERD refractory to PPI treatment.

After endoscopic confirmation of NERD, the probe based confocal endomicroscopy catheter will be inserted (CellVisio). The probe will be placed 5cm above the gastroesophageal junction (GEJ) defined as the top of gastric folds. Subsequently, 2.5cc of 10% fluorescein will be injected. The investigators will initiate a video recording of the microscopic images that is to start with the injection of the fluorescein and continue this video for 3 minutes. This video will be reviewed at a later time by 2 blinded endoscopists trained in confocal endomicroscopy interpretation. The goal is to see if the time to seeing fluorescein in the intracellular spaces correlates to response to therapy. The investigators will record time to first visualization of intrapapillary loops intracellular gaps, the time between visualization of intrapapillary loops and visualization of intracellular gaps in the entirety of the space between the loops. The investigators will also measurement of the general overall appearance. Having the recording of the microscopic images will allow a centralized reading time to each event and more accurate timing as the video can be stopped and reviewed in slow motion.

The investigators then will perform endomicroscopic assessment in four quadrants at 2cm, 5cm and 10cm above the gastroesophageal junction (GEJ). This will represent a single image acquisition video at each measurement with 4 separate views included. Computer analysis of the microscopic images will determine the average cell to cell junction distance, number of intrapapillary capillary loops, size of those intrapapillary capillary loops and overall saturation with fluorescein. Biopsies of the esophagus corresponding to the endomicroscopy sites will be collected for microscopic analysis.

Following endoscopy all patients will receive a 48h Bravo capsule or 24h impedance pH probe to quantitate acid and non-acid reflux events (if 24h probe used) . Standard calibration and insertion techniques provided by the manufacturer will be used. Standard symptom event recording for heartburn, regurgitation and non-cardiac chest pain will be used for the duration of the pH and impedance monitoring. A blinded investigator will interpret impedance and pH recording. The primary outcome will be the average Demeester Score.

For histopathology the specimen will be fixed in 10% formalin, embedded in paraffin and sectioned per standard clinical protocols. An expert pathologist will review pathology specimen for histological changes, specifically elongation of papillae, proliferation of basal cells, eosinophilic infiltration and dilated intercellular spaces.

Following their endoscopic evaluation, all patients will be randomized in a 1:1 ratio to receive either twice daily proton pump inhibitor (PPI) therapy for 8 weeks or sucralfate slurry 1g four times a day for 8 weeks. The patients will not be blinded to the treatment they receive. The patients will be contacted by phone to assess the symptoms, medication compliance and tolerance and to complete a RDQ and SF-36 at week 4. They will be seen in clinic 8 weeks as a follow-up visit and study wrap up. The 8 week visit is standard of care as that is how long the investigators typically follow patients with reflux symptoms. The investigators will also assess disease activity with a RDQ and SF-36 at this visit as well. Patients without adequate response to the medication will be offered cross over to the alternative medication with a 4 week phone assessment and 8 week clinic visit as described above. The investigators plan to enroll 40 patients at each site (total of 120 patients) and plan an interim analysis after the first 30 patients complete the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with reflux disease between the ages of 18 and 79 who have failed a trial of daily PPI.

Exclusion Criteria:

1. Barrett's esophagus
2. Use of high dose proton pump inhibitor within 4 weeks of study entry
3. Esophageal varices
4. Coagulopathy
5. GI cancer or mass
6. Previous surgery involving the esophagus, stomach or duodenum
7. Pregnancy
8. Allergy to either sucralfate or proton pump inhibitors

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Response to NERD treatment | 8 weeks
  We will use a validated measure of reflux disease - the reflux disease questionnaire (RDQ). This questionnaire consists of 12 items assessing various aspects of reflux disease. A score of more than 12 will be required for study entry. Response to treatment will be assessed based on reduction in scores on this survey.

SECONDARY OUTCOMES:
Confocal endomicroscopy findings | Immediate
  We will initiate a video recording of the microscopic images that is to start with the injection of the fluorescein and continue this video for 3 minutes. This video will be reviewed at a later time by 2 blinded endoscopists trained in confocal endomicroscopy interpretation.
Quality of life | 8 weeks
  We will use an SF-36 v2 survey to assess changes in quality of life at study entry and the finish of the study.

CONTACTS AND LOCATIONS:
Overall Officials: George B Smallfield, MD, MSPH, Principal Investigator — Virginia Commonwealth University
Locations (3):
- United States (3):
  - Ochsner Medical Center, Kenner, Louisiana
  - Medical University of South Carolina, Charleston, South Carolina
  - Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Background] Chu CL, Zhen YB, Lv GP, Li CQ, Li Z, Qi QQ, Gu XM, Yu T, Zhang TG, Zhou CJ, Rui-Ji, Li YQ. Microalterations of esophagus in patients with non-erosive reflux disease: in-vivo diagnosis by confocal laser endomicroscopy and its relationship with gastroesophageal reflux. Am J Gastroenterol. 2012 Jun;107(6):864-74. doi: 10.1038/ajg.2012.44. Epub 2012 Mar 13. PMID 22415199
- [Background] Law JD. Clinical and technical results from spinal stimulation for chronic pain of diverse pathophysiologies. Stereotact Funct Neurosurg. 1992;59(1-4):21-4. doi: 10.1159/000098912. PMID 1295042